CLINICAL TRIAL: NCT01221337
Title: Comparative Study of Two Haemodialyzers "VIE 2.1" Versus "EVODIAL2.2" in a Strategy of Heparin-free Haemodialysis (HFH)
Brief Title: Heparin Free Haemodialysis With Haemodialyzers "VIE" Versus "EVODIAL"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 10-PP-09
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Adult Chronic Haemodialysis Patients Since at Least 3 Months

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- haemodialyzer EVODIAL-haemodialyzer VIE (Other): Equal number of patients will start either with the haemodialyzer "VIE 2,1" or "EVODIAL 2,2" followed by a wash out period, before starting the other haemodialyzer.
  Interventions: Other: heparin free haemodialysis
- haemodialyzer VIE-haemodialyzer Evodial (Other): Equal number of patients will start either with the haemodialyzer "VIE 2,1" or "EVODIAL 2,2" followed by a wash out period, before starting the other haemodialyzer.
  Interventions: Other: heparin free haemodialysis

INTERVENTIONS:
Other: heparin free haemodialysis — Comparison of two haemodialyzers "VIE 2,1" versus "EVODIAL 2,2" in a strategy of heparin-free haemodialysis (HFH).

SUMMARY:
The adequate anti coagulation is an absolute necessity in order to avoid the extra-corporal circuit and haemodialyzer clotting and to perform an adequate renal replacement therapy during a haemodialysis session. In the cases of multiple coagulation defects having high haemorrhagic risk factors and the patients under anti-coagulation therapy, it is recommended to reduce the heparin doses or to do heparin free haemodialysis. Several strategies of low heparin or heparin free haemodialysis have been proposed till now, without a real success. The heparin coated polyacrylonitrile haemodialyser (EVODIAL) has been reported to have 90 % successful heparin-free haemodialysis sessions. On the other hand, the vitamin E coated polysulphone (VIE) has also been reported to have an anti oxidative and anti-thrombotic properties and a capacity to improve the haemorrheological factors of human blood, hence having a promising future to perform a successful haemodialysis session with less or without heparin. This randomised, multi-centric, cross-over and open study has been designed to compare non inferiority of the haemodialyzer VIE 2,1 versus EVODIAL2,2 with a risk alfa of 5% and an absolute accepted difference of 12 %.

ELIGIBILITY:
Inclusion Criteria:

-- Adult chronic haemodialysis patients since al least 3 months

* Two needles puncture of the fistula,
* Low molecular weight heparinization during haemodialysis sessions,
* Good fistula or central veinous catheter flow rate (blood pump flow rate ≥ 300 ml/min),
* Systolic blood pressure ≥ 110 mmHg (mean value of three last dialysis sessions.
* Patients capable to understand the design of the study and to follow the instructions
* Patients having the French social security system affiliation.

Non-inclusion criteria :

* C reactive protein > 30 mg/L.
* Single needle puncture of the fistula
* Active documented haemorrhage,
* Haemoglobin < 10 g/dl and/or need blood transfusion,
* Documented thrombophilia
* Patients waiting for renal graft
* Acute sepsis
* Fistula or catheter dysfunction
* Patients under anti-vitamine K
* Per dialytic hypotension requiring al least once a nurse intervention,
* Severe diseases (Dysglobulinemia, vascularitis, HIV…),
* Patients following another research protocol or have ended one less then one month before starting of this study.
* Pregnant or breast feeding patients,
* Minor patients or under law-protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The percentage of successful study periods with no circuit-clotting event leading to a premature interruption of any of the four dialysis sessions | during every haemodialysis sessions

SECONDARY OUTCOMES:
Duration of dialysis session without blood circuit clotting | during every haemodialysis sessions
Number of times saline rinsing has been required | during every haemodialysis
Degree of blood clots in the venous bubble trap | during every haemodialysis sessions
Quality of blood restitution | during every haemodialysis sessions
Dialysis adequacy (KT/V) | during every haemodialysis sessions
Haematological status | during every haemodialysis sessions
tolerance | during every haemodialysis sessions

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shariful ISLAM, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (2):
- France (2):
  - Centre Hospitalier, Avignon
  - CHU de Nice, Nice